CLINICAL TRIAL: NCT03719573
Title: Geriatric Assessment and Intervention in Older Patients Undergoing Surgery for Colorectal Cancer
Acronym: GEPOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Collaborators: Velux Fonden (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Troels Gammeltoft Dolin, MD, Principal Investigator, Department of internal Medicine, Herlev and Gentofte Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 123
Record Dates: First submitted 2018-10-19; First posted 2018-10-25 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Colon Cancer; Colon Neoplasm; Frail Elderly Syndrome; Colorectal Cancer
Keywords: Colon Cancer; Frailty; Geriatric assessment; perioperative care; exercise; quality of recovery; colorectal
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms; Frailty; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Physiotherapist assessing function status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Geriatric intervention (Experimental): A comprehensive geriatric assessment and intervention, including exercise program.
  Interventions: Other: Geriatric intervention
- control. (No Intervention): Usual treatment and care.

INTERVENTIONS:
Other: Geriatric intervention — A comprehensive geriatric assessment (CGA), focusing on co-morbidity, medication, cognitive status, depression, nutritional status and physical status is performed. The intervention is individualized according to the results of the CGA.
  Arms: Geriatric intervention

SUMMARY:
The GEPOC study investigates the effect of comprehensive geriatric assessment and intervention for frail older patients (65 years or older) undergoing elective surgery for colorectal cancer. the geriatric intervention will be pre- and postoperative. included in the intervention is an exercise intervention.

The main aim of the study us to see if the functional decline in this group can be reduced.

DETAILED DESCRIPTION:
This is a randomized, controlled trial on frail older patients (aged 65 years or older) with colorectal cancer. The patients will be randomized into two groups. The control group will receive standard surgical treatment. The intervention group will in addition go through a preoperative comprehensive geriatric assessment. The assessment will include evaluation of co-morbidity and medication, social status, nutritional status, cognition, depression and physical performance. This assessment will form basis of an individualized intervention. Patients in the intervention group will participate in planned exercise programs before surgery, perioperative and postoperative.

ELIGIBILITY:
Inclusion Criteria:

* elective surgery for colorectal cancer
* frail
* ability to read and speak danish (informed concent)

Exclusion Criteria:

* any physical condition that hinder physical exercise (eg. no legs)
* not able to concent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
30-second chair stand test (30s-CST) | baseline to 14 weeks after surgery
  functional test measuring lower body strength

SECONDARY OUTCOMES:
physical function and capacity - 6-minute-walk-test | baseline to 14 weeks after surgery
  6-minute-walk-test
physical function and capacity - hand grip strength | baseline to 14 weeks after surgery
  hand grip strength
physical function and capacity - 6-meter gait speed | baseline to 14 weeks after surgery
  6-meter gait speed
Patient reported Quality of Life: EORTC | baseline to 14 weeks after surgery
  EORTC European Organisation for Research and Treatment of Cancer questionnaire C30 (30-126 points where 30 is the worst)
Patient reported Quality of Life: EORTC ELD14 | baseline to 14 weeks after surgery
  EORTC European Organisation for Research and Treatment of Cancer questionnaire conjoined with ELD14 (Elderly Cancer Patient module) (14-54 points where 54 is the worst)
Quality of recovery after surgery: questionnaire | 1 day before surgery (baseline) to 3 days after surgery
  Measured with the questionnaire: Quality of Recovery - 15 questionnaire (0-150 points where 0 points is the worst)
body composition | baseline to 14 weeks after surgery.
  measured by Bioimpedance assessment
body composition | baseline to 14 weeks after surgery.
  measured by dual-energy x-ray absorptiometry
inflammatory biomarker - CRP | baseline to 14 weeks after surgery
  the concentration of CRP (CRP C-reactive Protein)
inflammatory biomarker - Interleukin 6 | baseline to 14 weeks after surgery
  the concentration of interleukin 6
inflammatory biomarker YKL-40 | baseline to 14 weeks after surgery
  the concentration of YKL-40 (YKL-40 is also known as Chitinase-3-like protein 1)
inflammatory biomarkers immuno-oncology | baseline to 14 weeks after surgery
  the concentration of 92 proteins associated with immuno-oncology (OLink)
sarcopenia biomarker GDF-11 | baseline to 14 weeks after surgery
  the concentration of GDF-11 (GDF Growth Differentiation Factor)
sarcopenia biomarker GDF | baseline to 14 weeks after surgery
  the concentration of GDF-15 (GDF Growth Differentiation Factor)
Postoperative complications | 30 days + 90 days
  Measured with Clavien Dindo classification (grade I-V where grade V is death)
readmission | 30 days after surgery and 90 days after surgery
  Number of patients being readmitted to hospital within 30 + 90 days after operation for colon surgery.
survival | 10 years
  number of survivors after surgery
mortality | baseline to 3 months
  number of patients death
number of patients to start up of adjuvant chemotherapy after surgery. | 14 weeks
  according to guidelines, if physical condition allows it (and patient accepts it).
start up time of adjuvant chemotherapy after surgery | 14 weeks
  measured in days (if relevant)
number of series of adjuvant chemotherapy | 14 weeks
doses of adjuvant chemotherapy | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Julia S Johansen, MD, PhD, Study Chair — Professor
Locations (1):
- Herlev and Gentofte Hospital, Herlev, Region H, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
TBA

REFERENCES:
- [Derived] Dolin TG, Mikkelsen MK, Jakobsen HL, Vinther A, Zerahn B, Nielsen DL, Johansen JS, Lund CM, Suetta C. The prevalence of sarcopenia and cachexia in older patients with localized colorectal cancer. J Geriatr Oncol. 2023 Jan;14(1):101402. doi: 10.1016/j.jgo.2022.11.001. Epub 2022 Nov 21. PMID 36424269
- [Derived] Dolin TG, Mikkelsen M, Jakobsen HL, Nordentoft T, Pedersen TS, Vinther A, Zerahn B, Vistisen KK, Suetta C, Nielsen D, Johansen JS, Lund CM. Geriatric assessment and intervention in older vulnerable patients undergoing surgery for colorectal cancer: a protocol for a randomised controlled trial (GEPOC trial). BMC Geriatr. 2021 Jan 30;21(1):88. doi: 10.1186/s12877-021-02045-9. PMID 33516195